CLINICAL TRIAL: NCT02563951
Title: A Phase I Pharmacokinetic Study of Granisetron Hydrochloride Nasal Spray (GNS) in Healthy Volunteers
Brief Title: Study of Granisetron Hydrochloride Nasal Spray (GNS) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maxinase Life Sciences Ltd. (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNS-CL001
Record Dates: First submitted 2015-09-16; First posted 2015-09-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: Nausea; Vomiting; Chemotherapy; Radiation therapy
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting | interventions — Granisetron; Injections, Intravenous; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- GNS Spray 0.5mg (Experimental): One spray of GNS 0.5mg/spray into right nostril.
  Interventions: Drug: GNS Spray 0.5mg
- GNS Spray 1.0mg (Experimental): One spray of GNS 0.5mg/spray into both left and right nostril.
  Interventions: Drug: GNS Spray 1.0mg
- GNS Spray 2.0mg (Experimental): One spray of GNS 1.0mg/spray into both left and right nostril.
  Interventions: Drug: GNS Spray 2.0mg
- Kytril 1mg (IV injection) (Active Comparator): A dose of 1mg of Granisetron IV injection (kytril 1mL, 3mg/mL/vial) will be administered as a slow IV injection (over 30 seconds)
  Interventions: Drug: Kytril 1mg (IV injection)
- Kytril 1mg (Tablet) (Active Comparator): a single dose (kytril 1mg, one tablet) orally administered with 240mL of water
  Interventions: Drug: Kytril 1mg (Tablet)

INTERVENTIONS:
Drug: GNS Spray 0.5mg
  Other Names: Granisetron Nasal Spray
  Arms: GNS Spray 0.5mg
Drug: GNS Spray 1.0mg
  Other Names: Granisetron Nasal Spray
  Arms: GNS Spray 1.0mg
Drug: GNS Spray 2.0mg
  Other Names: Granisetron Nasal Spray
  Arms: GNS Spray 2.0mg
Drug: Kytril 1mg (IV injection)
  Other Names: Granisetron
  Arms: Kytril 1mg (IV injection)
Drug: Kytril 1mg (Tablet)
  Other Names: Granisetron
  Arms: Kytril 1mg (Tablet)

SUMMARY:
The purpose of this study is to examine the pharmacokinetics (PK), safety and tolerability of 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of Granisetron Hydrochloride Nasal Sprays (GNS) as compared to Granisetron IV Injection and Granisetron Tablet in healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between the ages of 20-64 years
2. Body Mass Index (BMI) of 18.5 (inclusive) to 24 kg/m2; and a total body weight >45 kg
3. Accessible vein for blood sampling
4. No significant abnormalities in electrocardiogram (ECG) recording as per sites' local practice
5. No significant abnormalities in general physical examination as per sites' local practice
6. No significantly abnormal findings in laboratory assessments including hematology, biochemistry and urinalysis as per site's local practice
7. A signed and dated written informed consent must be obtained from the subject prior to study participation
8. Capable of understanding and willing to comply with study procedures
9. A negative serum pregnancy test before the first dose of study drug must be available for women of childbearing potential

Exclusion Criteria:

1. Females who are pregnant, breast-feeding or have positive pregnancy test
2. History of hypersensitivity to granisetron or its analogs
3. Subjects with nasal ulcer, septal perforation, or other nasal conditions that may interfere with nasal administration and determined by the investigator to be ineligible
4. Subjects with a QT interval greater than 500 ms or with acute ischemic changes or cardiac abnormality predisposing to arrhythmia on screening electrocardiogram (ECG) or by history
5. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or other significant disease or clinical findings at screening and determined by the investigator to be ineligible
6. Subjects with a history of drug and/or alcohol abuse within 12 months prior to dosing
7. Inability to read and/or sign the consent form
8. Treatment with any other investigational drug during the 4 weeks prior to the initial dosing for this study
9. Subjects who have donated or lost more than 250 ml blood within 2 months prior to the initial dosing for this study
10. Male and female subjects with reproductive potential who are not willing to use effective method of contraception. Use of hormonal contraceptive is not allowed during the study period
11. Clinical significant rhinitis or rhinorrhea at screening determined by the investigator to be ineligible
12. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to dosing of study medication
13. For subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums, etc.), 2 weeks abstinence is required
14. Conditions upon screening which might contraindicate or require that caution be used in the administration of granisetron

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PK Parameter: Area under the plasma concentration-time curve from zero (0) hours to infinity (∞) (AUC(0-∞)) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of GNS and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: Area under the plasma concentration-time curve from zero (0) hours to last quantifiable concentration(t) (AUC(0-t)) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of GNS and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: Peak Plasma Concentration (Cmax) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of GNS and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: Area under the plasma concentration-time curve from zero (0) hours to infinity (∞) (AUC(0-∞)) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
PK Parameter: Area under the plasma concentration-time curve from zero (0) hours to last quantifiable concentration (t) (AUC(0-t)) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
PK Parameter: Peak Plasma Concentration (Cmax) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose

SECONDARY OUTCOMES:
PK Parameter: Time to maximum plasma concentration (Tmax) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of Granisetron Hydrochloride Nasal Sprays (GNS) and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: Time to maximum plasma concentration (Tmax) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
PK Parameter: elimination constant rate (Kel) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of Granisetron Hydrochloride Nasal Sprays (GNS) and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: elimination constant rate (Kel) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
PK Parameter: half-life (t1/2) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of Granisetron Hydrochloride Nasal Sprays (GNS) and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: half-life (t1/2) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
PK Parameter: absolute bioavailability (F) for 3 intranasal (IN) doses (0.5, 1.0 and 2.0 mg) of Granisetron Hydrochloride Nasal Sprays (GNS) and Granisetron IV Injection | within 1 hour prior to drug administration; 5, 10, 15, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
PK Parameter: absolute bioavailability (F) for Granisetron Tablet | within 1 hour prior to drug administration; 15, 30, 45 minutes, and 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours post-dose
Report adverse events and measure vital signs over trial period. | These will be measured from 30 mins pre-dose to every 3 hours until 12 hours post-dose, then at 24 and 36 hours post-dose
12-Lead ECG assessment | This will be measured at screening, and 24, 36 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Min Chu, M.D Ph.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Neihu District, Taipei City, Taiwan